CLINICAL TRIAL: NCT02621424
Title: Repetitive Transcranial Magnetic Stimulation for Dementia
Acronym: rTMS for demen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E1889-P; RX14-009 (Other Grant/Funding Number: VA)
Record Dates: First submitted 2015-11-23; First posted 2015-12-03 (Estimated); Results first posted 2020-05-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Dementia; Mild Cognitive Impairment
Keywords: dementia; Mild Cognitive Impairment (MCI); RTMS; CVLT
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- RTMS (Experimental): repetitive transcranial magnetic stimulation
  Interventions: Device: RTMS
- sham (Sham Comparator): sham noise to block the sound of treatment
  Interventions: Device: sham

INTERVENTIONS:
Device: RTMS — stimulation of the brain with magnetic pulses
  Arms: RTMS
Device: sham — sham noise to block the sound of stimulation
  Arms: sham

SUMMARY:
The purpose is to is to study if repetitive transcranial magnetic stimulation (rTMS) improves cognitive function in patients with neurodegenerative conditions which may manifest as mild to moderate cognitive impairment and, in late phase, dementia. This study also intends to investigate if the responses to rTMS intervention are either positively or negatively correlated with the initial severity of cognitive impairment.

DETAILED DESCRIPTION:
The primary hypothesis is that rTMS applied to the dorsolateral prefrontal cortex will lead to improved memory, language and executive function compared to patients who receive a sham, control treatment. The improvement is defined as having higher performance on the California Verbal Learning Test (CVLT-II). Secondary Hypotheses are that:

* 1: rTMS- will lead to higher performance on secondary cognitive measures relating to executive function and naming compared to performance by participants in the sham treatment group at the termination of treatment; and that
* 2: rTMS-induced memory improvement parallels changes in serum and cerebrospinal fluid (CSF) brain-derived neurotrophic factor (BDNF) levels after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Veterans aged 55 years or older
* Diagnosed with Mild Cognitive Impairment (MCI) or dementia likely due to Alzheimer's disease.
* Ability to obtain a Motor Threshold, determined during the screening process.
* With an adequately stable condition and living environment to enable attendance at scheduled clinic visits.
* If on a prescription medication for cognition that medication dose will be stable for at least 4 weeks prior to randomization into the study and participant will be willing to remain on a stable regimen during the acute treatment phase.
* Able to read, verbalize understanding, and voluntarily sign the Informed Consent Form to be signed by the participant, or a designated legal representative when the participant lacks decision making capacity prior to participating in any study- specific procedures or assessments.

Exclusion Criteria:

* Patients with prior exposure to rTMS or electroconvulsive therapy (ECT).
* Unable to safely withdraw, at least two weeks prior to treatment commencement, from medications that substantially increase the risk of having seizures.
* Have a cardiac pacemaker or a cochlear implant.
* Have an implanted device deep brain stimulation or metal in the brain
* Current substance abuse not including caffeine or nicotine as determined by patient report or chart review.
* Active current suicidal intent or plan as determined by patient report or chart review.
* Current or Prior history of a seizure disorder as determined by patient report or chart review
* Traumatic brain injury within the last two months
* Participation in another concurrent interventional clinical trial
* Known current psychosis as determined by patient report or chart review.
* Current or prior history of a mass lesion, cerebral infarct or other non-cognitive, active central nervous system (CNS) disease that would increase the risk for seizure.
* Not fluent in English or a hearing impairment severe enough to impair comprehension

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2025-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jauhtai J Cheng, MD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng J, Fairchild JK, McNerney MW, Noda A, Ashford JW, Suppes T, Chao SZ, Taylor J, Rosen AC, Durazzo TC, Lazzeroni LC, Yesavage J. Repetitive Transcranial Magnetic Stimulation as a Treatment for Veterans with Cognitive Impairment and Multiple Comorbidities. J Alzheimers Dis. 2022;85(4):1593-1600. doi: 10.3233/JAD-210349. PMID 34958013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two hundred and twenty nine patients were screened. 43 patients signed consent. 32 were enrolled.
Pre-assignment Details: Thirty two patients were enrolled.
Period: Overall Study
Arm/Group | RTMS | Sham
Started | 14 | 18
Completed | 13 | 16
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RTMS | Sham | Total
Number analyzed (Participants) | 14 | 18 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (7.4) | 70.4 (7.7) | 70.8 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 14 | 17 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 0 | 2 | 2
  White | 10 | 12 | 22
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 18 | 32
neuropsychological testing [Count of Participants; unit: Participants] | 14 | 18 | 32

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline CVLT Scores After Treatment and 4 Month Later
Description: Changes of California verbal learning test scores (CVLT) from baseline after treatment and 4 months later.
  CVLT is 16 points scoring system. (minimum=0, maximum=16, higher the better memory).
Time Frame: Assessed at baseline, end of treatment, and 4-month post-treatment follow up
Population: Sham arm: 18 started, 2 withdrew, 3 did not test properly at baseline, 1 did not show for follow up.
  13 sets of data were available at baseline, 13 sets were available at end of treatment, 12 sets were available at follow up. Active arm: 14 started, one withdrew, one did not show for follow up. 13 sets of data were available at baseline, 13 sets were available at end of treatment, 12 sets were available at follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTMS | Sham
Number analyzed (Participants) | 13 | 13
score on a scale
  Baseline | 8.5 (4.6) | 9.4 (3.8)
  End of treatment | 8.6 (4.3) | 8.3 (3.7)
  4 month follow up: number analyzed (Participants) | 12 | 12
  4 month follow up | 10.1 (4.1) | 9.2 (4.2)

2. Secondary Outcome: Changes in Boston Naming After Treatment
Description: Changes in Boston Naming Test (BNT) from baseline was analyzed. BNT is a 60 points scoring system. (minimum=0, maximum=60, higher the better).
Time Frame: Assessed at baseline, end of treatment, and 4-month post-treatment follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RTMS | Sham
Number analyzed (Participants) | 13 | 13
units on a scale
  baseline | 52.7 (12.4) | 53.7 (8.3)
  End of treatment | 52.8 (13.2) | 56.5 (3.6)
  4 month followup: number analyzed (Participants) | 12 | 12
  4 month followup | 54.4 (13.1) | 55.0 (5.3)

3. Secondary Outcome: Changes in Plasma BDNF Levels After Treatment
Description: Changes in BDNF plasma levels (pg/ml) from baseline were analyzed after treatment.
  BDNF is a plasma biomarker, minimum=0, no maximum. Higher number means more BDNF synthesis).
Time Frame: within a week following the last treatment session and 4 months later
Population: Sham arm: 18 started, 13 had baseline BDNF collected, two withdrew. 13 sets of data were available at baseline, 11 sets of data were available at end of treatment. Active arm: 14 started, two did not have BDNF collected. 12 sets of data were available at baseline and at end of treatment.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | RTMS | Sham
Number analyzed (Participants) | 12 | 13
pg/ml
  baseline | 5089 (3508) | 5054 (3440)
  post treatment: number analyzed (Participants) | 12 | 11
  post treatment | 5229 (3713) | 5350 (4981)

4. Secondary Outcome: Changes in Animal Fluency After Treatment and 4 Months Later
Description: Animal Fluency (AF) is a scoring system to assess the ability to generate a list of related words.
  The score is the number of animals the examinee can name in one minute time. (Minimum = 0, No maximum, higher the better).
Time Frame: Assessed at baseline, end of treatment, and 4-month post-treatment follow up
Population: Sham arm: 18 started, 2 withdrew, 3 did not test properly at baseline, 1 did not show for follow up.
  13 sets of data were available at baseline, 13 sets were available at end of treatment, 12 sets were available at follow up. Active arm: 14 started, one withdrew, one did not test properly at end of treatment, one did not show for follow up.
  13 sets of data were available at baseline, 12 sets were available at end of treatment, 12 sets were available at follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RTMS | Sham
Number analyzed (Participants) | 13 | 13
units on a scale
  baseline | 17.8 (6.6) | 15.8 (3.4)
  end of treatment: number analyzed (Participants) | 12 | 13
  end of treatment | 15.6 (4.9) | 16.8 (3.0)
  4 month followup: number analyzed (Participants) | 12 | 12
  4 month followup | 15.8 (5.4) | 16.9 (5.1)

5. Secondary Outcome: Changes in Trail Making B Test Score After Treatment and 4 Months Later
Description: Trail making B is a scoring system for the assessment of the mental flexibility, processing speed and executive function. The score is the time (in seconds) it takes for the examinee to draw line segments connecting sequentially from 1-A-2-B-3....all the way to12-L-13. (The lower score means faster speed and means better performance. The minimum is (hypothetically) zero. There is no maximum. However, in some test centers, the maximum allowed time is 200 seconds.
Time Frame: Assessed at baseline, end of treatment, and 4-month post-treatment follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | RTMS | Sham
Number analyzed (Participants) | 13 | 13
Seconds
  baseline | 187.5 (222.2) | 172.8 (94.8)
  end of treatment | 179.8 (207.7) | 150.4 (64.9)
  4 month followup: number analyzed (Participants) | 12 | 12
  4 month followup | 185.8 (237.8) | 197.6 (204.9)

6. Secondary Outcome: Brief Visual Memory Test (BVMT)
Description: A piece of paper with 6 simple drawings is presented to the subject for 10 seconds. The subject is then asked to draw these drawings from memory. The process is repeated three times to assess visual memory and learning. Each correct drawing scores two pints. Maximum score for three trials is 36. Minimum score is 0. Higher the better.
Time Frame: assessed at baseline, end of treatment and 4-month post-treatment follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTMS | Sham
Number analyzed (Participants) | 13 | 13
score on a scale
  Baseline | 18.9 (9.0) | 17.4 (6.4)
  End of treatment | 19.4 (8.7) | 17.2 (7.3)
  4 month follow up: number analyzed (Participants) | 12 | 12
  4 month follow up | 18.8 (7.5) | 16.6 (7.0)

7. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: MoCA is a one page, 30 point cognitive screening test. It test the following cognitive domains:
  1. short-term memory (5 points)- two learning trials of five nouns and delayed recall after approximately five minutes.
  2. visuospatial abilities - clock-drawing task (3 points) and copy a cube (1 point).
  3. executive functions - alternation task abbreviated trail-making B (1 point), and a two-item verbal abstraction task (2 points).
  4. attention, concentration, and working memory - a sustained attention task (target detection using tapping; 1 point), a serial subtraction task (3 points), and digits forward and backward (1 point each).
  5. language - three-item confrontation naming (3 points), repetition of two sentences (2 points), and verbal fluency (1 point).
  6. abstract reasoning - describe the similarity of tasks (2 points).
  7. orientation to time and place (6 points). Minimum score: 0. Maximum score: 30. Higher the better.
Time Frame: Assessed at baseline, end of treatment, and 4-month post-treatment follow up
Population: Sham arm: 18 started, 2 withdrew, 3 did not test properly at baseline, 1 did not show for follow up.
  13 sets of data were available at baseline, 13 sets were available at end of treatment, 12 sets were available at follow up. Active arm: 14 started, one withdrew, two did not test properly at end of treatment, one did not show for follow up.
  13 sets of data were available at baseline, 11 sets were available at end of treatment, 12 sets were available at follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RTMS | Sham
Number analyzed (Participants) | 13 | 13
score on a scale
  baseline | 22.4 (6.1) | 24.3 (3.0)
  end of treatment: number analyzed (Participants) | 11 | 13
  end of treatment | 22.0 (6.0) | 24.1 (3.9)
  4 month follow up: number analyzed (Participants) | 12 | 12
  4 month follow up | 24.8 (6.2) | 24.7 (4.4)

ADVERSE EVENTS:
Time Frame: 1 year post treartment
Groups:
- RTMS: repetitive transcranial magnetic stimulation
  mild headache and irritation at the site of stimulation were reported and thought to be treatment-related. These event were mild and only lasted a day or two.
  There were other reported events and were reviewed with the IRB. They were determined to be not related to RTMS treatment.
- Sham: sham noise to block the sound of treatment Low amplitude electrical stimulation was used to simulate the sensation of RTMS. The electrical stimulation to the scalp can cause mild sense of irritation, which only occurs when the stimulation is turned on.
  There were other reported events and were reviewed with the IRB. They were determined to be not related to RTMS treatment.
Arm/Group | RTMS | Sham
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/14 | 2/18
Other Adverse Events (participants affected / at risk) | 0/14 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RTMS (N=14) | Sham (N=18)
epilepsy (Nervous system disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/24/NCT02621424/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/24/NCT02621424/SAP_001.pdf
  • Informed Consent Form (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT02621424/ICF_002.pdf